CLINICAL TRIAL: NCT03541200
Title: An Open-label, Long Term Extension Study of MT-8554 in Postmenopausal Women Experiencing Moderate to Severe Vasomotor Symptoms Who Completed Study MT-8554-A01
Brief Title: Long-term Safety and Efficacy Study of MT-8554 in Postmenopausal Women With Vasomotor Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-8554-A02
Record Dates: First submitted 2018-03-29; First posted 2018-05-30 (Actual); Results first posted 2022-10-03 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Vasomotor Symptoms (VMS)

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label (Experimental): MT-8554
  Interventions: Drug: MT-8554

INTERVENTIONS:
Drug: MT-8554 — MT-8554 Oral

SUMMARY:
An open-label, long term extension study of MT-8554 in postmenopausal women experiencing moderate to severe vasomotor symptoms who completed Study MT-8554-A01

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent to participate in this study.
* Subjects who complete the preceding trial (Study MT-8554-A01) through Week 12.

Exclusion Criteria:

* Subjects who meet the withdrawal criteria for the proceeding trial (Study MT-8554-A01)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Head of Medical Science, Study Director — Tanabe Pharma America, Inc.
Locations (49):
- United States (49):
  - Research Site, Birmingham, Alabama
  - Research Site, Dothan, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Norwalk, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Denver, Colorado
  - Research Site, New London, Connecticut
  - Research Site, Clearwater, Florida
  - Research Site, Crystal River, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Jupiter, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Ponte Vedra, Florida
  - Research Site, Port Saint Lucie, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Wellington, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Sandy Springs, Georgia
  - Research Site, Idaho Falls, Idaho
  - Research Site, Hutchinson, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Marrero, Louisiana
  - Research Site, Metairie, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Kalamazoo, Michigan
  - Research Site, Saginaw, Michigan
  - Research Site, Kansas City, Missouri
  - Research Site, Missoula, Montana
  - Research Site, Las Vegas, Nevada
  - Research Site, Lawrenceville, New Jersey
  - Research Site, Morehead City, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Englewood, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Bristol, Tennessee
  - Research Site, Jackson, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Fort Worth, Texas
  - Research Site, Schertz, Texas
  - Research Site, Draper, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Norfolk, Virginia
  - Research Site, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- MT-8554: MT-8554 10mg QD for 52 weeks, followed MT-8554 1mg or 5mg or 10mg or placebo QD for 12 weeks in MT-8554-A01 study. Based upon the results of MT-8554-A01 study, the dose was changed from 10 mg to 5 mg during the study.
Period: Overall Study
Arm/Group | MT-8554
Started | 190
Completed | 77
Not Completed | 113
Not completed — Adverse Event | 19
Not completed — Death | 1
Not completed — Lost to Follow-up | 10
Not completed — Physician Decision | 1
Not completed — Protocol Violation | 51
Not completed — Withdrawal by Subject | 23
Not completed — other | 8

BASELINE CHARACTERISTICS:
Population: 3 subjects did not take any study medication so these subjects were excluded from the Safety Population.
Arm/Group | MT-8554
Number analyzed (Participants) | 187
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (6.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 187
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 47
  White | 138
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Adverse Events
Time Frame: 52 Weeks
Population: 3 subjects did not take any study medication so these subjects were excluded from the Safety Population.
Measure: Number; unit: percentage of subjects
Arm/Group | MT-8554
Number analyzed (Participants) | 187
percentage of subjects | 56.7

2. Primary Outcome: Percentage of Subjects With Serious Adverse Events
Time Frame: 52 Weeks
Population: 3 subjects did not take any study medication so these subjects were excluded from the Safety Population.
Measure: Number; unit: percentage of subjects
Arm/Group | MT-8554
Number analyzed (Participants) | 187
percentage of subjects | 3.2

3. Primary Outcome: Percentage of Subjects With Clinical Laboratory Tests Abnormalities
Description: Hematology, biochemistry, coagulation and urinalysis
Time Frame: 52 Weeks
Population: 3 subjects did not take any study medication so these subjects were excluded from the Safety Population.
Measure: Number; unit: percentage of subjects
Arm/Group | MT-8554
Number analyzed (Participants) | 187
percentage of subjects | 15.5

4. Primary Outcome: Change in Blood Pressure
Description: Systolic and diastolic blood pressure
Time Frame: Baseline and 52 Weeks
Population: 3 subjects did not take any study medication so these subjects were excluded from the Safety Population. The number of subjects with SBP and DBP results at Week 52 are mentioned in each row "number of participants analyzed".
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MT-8554
Number analyzed (Participants) | 187
mmHg
  Systolic Blood Pressure: number analyzed (Participants) | 158
  Systolic Blood Pressure | 1.3 (11.36)
  Diastolic Blood Pressure: number analyzed (Participants) | 158
  Diastolic Blood Pressure | -0.4 (7.65)

5. Primary Outcome: Change in Heart Rate
Time Frame: Baseline and 52 Weeks
Population: 3 subjects did not take any study medication so these subjects were excluded from the Safety Population. The number of subjects with heart rate result at Week 52 are mentioned in row "number of participants analyzed".
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | MT-8554
Number analyzed (Participants) | 156
beats/min | 2.6 (7.96)

6. Primary Outcome: Change in ECG Parameters
Description: PR, QRS, QT and QTc
Time Frame: Baseline and 52 Weeks
Population: 3 subjects did not take any study medication so these subjects were excluded from the Safety Population. The number of subjects with each parameter result at Week 52 are mentioned in each row "number of participants analyzed".
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | MT-8554
Number analyzed (Participants) | 187
msec
  PR: number analyzed (Participants) | 155
  PR | 0.4 (16.34)
  QRS: number analyzed (Participants) | 156
  QRS | -0.2 (9.46)
  QT: number analyzed (Participants) | 156
  QT | -6.8 (22.86)
  QTcF: number analyzed (Participants) | 151
  QTcF | -0.6 (18.60)
  QTcB: number analyzed (Participants) | 154
  QTcB | 1.2 (19.66)

7. Primary Outcome: Change in Endometrial Thickness as Measured by Transvaginal Ultrasound
Time Frame: Baseline and 52 Weeks
Population: 3 subjects did not take any study medication so these subjects were excluded from the Safety Population. The number of subjects with endometrial thickness result at Week 52 are mentioned in row "number of participants analyzed".
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | MT-8554
Number analyzed (Participants) | 34
mm | -0.138 (1.4765)

8. Primary Outcome: Percentage of Participants With Endometrial Hyperplasia as Measured by Endometrial Biopsy
Time Frame: 52 Weeks
Population: 3 subjects did not take any study medication so these subjects were excluded from the Safety Population.
Measure: Number; unit: percentage of subjects
Arm/Group | MT-8554
Number analyzed (Participants) | 187
percentage of subjects | 0

9. Secondary Outcome: Change in Average Daily Frequency of Moderate to Severe VMS
Description: Subjects were asked to record frequency and severity of VMS in an electronic diary. Severity levels are defined as follows.
  Mild : Sensation of heat without sweating
  Moderate : Sensation of heat with sweating, able to continue activity
  Severe : Sensation of heat with sweating, causing cessation of activity
Time Frame: Baseline and 52 Weeks
Population: 6 subjects did not have any post-baseline efficacy assessment so these subjects were excluded from the Intent-to-treat population.The number of subjects with VMS frequency result at Week 52 are mentioned in row "number of participants analyzed".
Measure: Mean (Standard Deviation); unit: episodes/day
Arm/Group | MT-8554
Number analyzed (Participants) | 64
episodes/day | -2.71 (4.974)

10. Secondary Outcome: Change in Average Daily Severity Score of Mild to Severe VMS
Description: Baseline VMS severity score : (1xFmi + 2xFmo + 3xFse)/(Fmi + Fmo + Fse)
  VMS severity score for a specific week during the open label treatment period :(1xFmi+2xFmo+3xFse)/(Fmi+Fmo+Fse)
  Fmi, Fmo, and Fse are the daily frequencies of mild, moderate, and severe VMS respectively.
  The severity score of VMS ranged from 0 (lowest severity) to 3 (highest severity).
Time Frame: Baseline and 52 Weeks
Population: 6 subjects did not have any post-baseline efficacy assessment so these subjects were excluded from the Intent-to-treat population.The number of subjects with VMS severity result at Week 52 are mentioned in row "number of participants analyzed".
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MT-8554
Number analyzed (Participants) | 64
units on a scale | -0.325 (0.6804)

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: 3 subjects did not take any study medication so these subjects were excluded from the Safety Population.
Arm/Group | MT-8554
All-Cause Mortality (participants affected / at risk) | 1/187
Serious Adverse Events (participants affected / at risk) | 6/187
Other Adverse Events (participants affected / at risk) | 91/187
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MT-8554 (N=187)
Diverticulitis (Infections and infestations) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cystocele (Reproductive system and breast disorders) | 1
Rectocele (Reproductive system and breast disorders) | 1
Vaginal prolapse (Reproductive system and breast disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MT-8554 (N=187)
Diarrhoea (Gastrointestinal disorders) | 2
Diverticulum (Gastrointestinal disorders) | 3
Gastritis (Gastrointestinal disorders) | 2
Hypoaesthesia oral (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 3
Paraesthesia oral (Gastrointestinal disorders) | 14
Vomiting (Gastrointestinal disorders) | 3
Chills (General disorders) | 2
Fatigue (General disorders) | 2
Feeling cold (General disorders) | 4
Feeling hot (General disorders) | 9
Bacterial vaginosis (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 3
Influenza (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 10
Urinary tract infection (Infections and infestations) | 7
Viral upper respiratory tract infection (Infections and infestations) | 2
Accidental overdose (Injury, poisoning and procedural complications) | 4
Overdose (Injury, poisoning and procedural complications) | 5
Activated partial thromboplastin time prolonged (Investigations) | 3
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 3
Blood cholesterol increased (Investigations) | 3
Blood creatine phosphokinase increased (Investigations) | 3
Blood pressure increased (Investigations) | 2
Blood triglycerides increased (Investigations) | 3
Body temperature decreased (Investigations) | 2
Electrocardiogram abnormal (Investigations) | 2
Gamma-glutamyltransferase increased (Investigations) | 4
International normalised ratio increased (Investigations) | 4
Prothrombin time prolonged (Investigations) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 6
Burning sensation (Nervous system disorders) | 2
Headache (Nervous system disorders) | 3
Hypoaesthesia (Nervous system disorders) | 8
Hypogeusia (Nervous system disorders) | 2
Migraine (Nervous system disorders) | 3
Paraesthesia (Nervous system disorders) | 14
Sciatica (Nervous system disorders) | 2
Depression (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 5
Vaginal haemorrhage (Reproductive system and breast disorders) | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Flushing (Vascular disorders) | 2
Hot flush (Vascular disorders) | 2
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-08-13): https://cdn.clinicaltrials.gov/large-docs/00/NCT03541200/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/00/NCT03541200/SAP_001.pdf